CLINICAL TRIAL: NCT04503304
Title: Effect of Hip Abductors Versus Knee Extensor Strengthening on Pain,Function and Quadriceps Isometric Strength in Knee Osteoarthritis
Brief Title: Effect of Hip Abductors Versus Knee Extensor Strengthening in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aalaa Mohamed El-Amin Sweelam, Teaching Assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hip Abductors strength in KOA
Record Dates: First submitted 2020-08-01; First posted 2020-08-07 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis AND Hip Abductors AND Quadriceps
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: 2 groups; hip abductors strengthening (HAS) group a will receive hip abductors strengthening exercises, and knee extensors strengthening (KES) group will receive quadriceps strengthening exercise.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HAS group (Experimental): hip abductors strengthening group
  1. Hip abduction -standing[Ferber et al.,2015].
  2. Sidelying hip abduction(clamshell)[Schache et al.,2016].
  3. lateral leg raise: in brief, the patients lie down on bed on the unaffected side, with the resistance band positioned around the distal thigh of the affected limb.;later, they raise the above lower limbs upwards for about 30 degrees, stay for 5- 10 s and slowly lay down[Xie et al.,2018].
  4. pelvic lift training, specifically, patients stand single-leg off the side at a 10-cm step. Later, they begin with the other limb that is lower than the step level, and contract the stance-limb hip abductor to raise the free leg to the step level while keeping the stance knee extended[Xie et al.,2018].
  5. Stretching Hamstrings [Fukuda et al.,2012]. Number of sets = 3, Repetitions =10 repetitions for each set
  Interventions: Other: Exercises
- KES group (Active Comparator): knee extensors strengthening group
  1. Isometric quadriceps setting
  2. Knee extensions from sitting with knee bend to 90
  3. Terminal knee extension from sitting.
  4. Stretching Hamstrings Number of sets = 3, Repetitions =10 repetitions for each set
  Interventions: Other: Exercises

INTERVENTIONS:
Other: Exercises — already included in arm/group descriptions.

SUMMARY:
This study will try to answer the following question:

Would strengthening of hip abductors be equal to, or more effective than, knee extensors strengthening in improving pain, function and knee extensors isometric strength in patients with knee Osteoarthritis

DETAILED DESCRIPTION:
A total of 70 patients with knee Osteoarthritis will be recruited All patients who will participate in the study will be referred by orthopedists. Patients with knee osteoarthritis will be included with age ranges from 50-70. They will be randomized into 2 groups; hip abductors strengthening (HAS) group a will receive hip abductors strengthening exercises, and knee extensors strengthening (KES) group will receive quadriceps strengthening exercise.

All patients who will meet the study criteria will get a complete knowledge of the objectives and procedures of the study.

Inclusion criteria:

1. Patients with knee Osteoarthritis grade II- III Kellgren- Lawrence scores
2. Their age is 50-70[Wang et al.,2019].
3. Body mass index (BMI) 25-30.

Exclusion criteria:

1. Patients who had surgical intervention in the knee and/or hip.
2. Fracture in the lower limbs.
3. Malignancy
4. Any associated ligamentous injuries in knee or ankle.
5. Spinal Cord Injury.
6. Hormonal imbalance or on hormonal therapy
7. Knee injection within the last 6 months prior to the study. Outcome parameters including Quadriceps Muscle Strength, the arabic version of Western Ontario and McMaster Universities Arthritis Index questionnaire total score and 3 subscales and Timed Up and Go test score

ELIGIBILITY:
Inclusion Criteria:

1. Patients with knee OA grade II- III Kellgren- Lawrence scores
2. Their age is 50-70[Wang et al.,2019].
3. Body mass index (BMI) 25-30.

Exclusion Criteria:

1. Patients who had surgical intervention in the knee and/or hip.
2. Fracture in the lower limbs.
3. Malignancy
4. Any associated ligamentous injuries in knee or ankle.
5. Spinal Cord Injury.
6. Hormonal imbalance or on hormonal therapy
7. Knee injection within the last 6 months prior to the study.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Quadriceps Muscle Strength assessment | 6 weeks
  Quadriceps Muscle Strength assessment using Hand held Dynamometer
lower limb functional disability | 6 weeks
  Measuring lower limb functional disability using The Arabic version of reduced WOMAC (ArWOMAC) index
Knee function | 6 weeks
  Measuring function using The Timed Up & Go Test (TUG):

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
protocol copy, informed consent, statistical analysis
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Alghadir A, Anwer S, Brismee JM. The reliability and minimal detectable change of Timed Up and Go test in individuals with grade 1-3 knee osteoarthritis. BMC Musculoskelet Disord. 2015 Jul 30;16:174. doi: 10.1186/s12891-015-0637-8. PMID 26223312
- [Background] Alghadir A, Anwer S, Iqbal ZA, Alsanawi HA. Cross-cultural adaptation, reliability and validity of the Arabic version of the reduced Western Ontario and McMaster Universities Osteoarthritis index in patients with knee osteoarthritis. Disabil Rehabil. 2016;38(7):689-94. doi: 10.3109/09638288.2015.1055380. Epub 2015 Jun 11. PMID 26066566
- [Background] Alnahdi AH, Zeni JA, Snyder-Mackler L. Hip abductor strength reliability and association with physical function after unilateral total knee arthroplasty: a cross-sectional study. Phys Ther. 2014 Aug;94(8):1154-62. doi: 10.2522/ptj.20130335. Epub 2014 Mar 20. PMID 24652473
- [Background] Altman R, Alarcon G, Appelrouth D, Bloch D, Borenstein D, Brandt K, Brown C, Cooke TD, Daniel W, Gray R, et al. The American College of Rheumatology criteria for the classification and reporting of osteoarthritis of the hand. Arthritis Rheum. 1990 Nov;33(11):1601-10. doi: 10.1002/art.1780331101. PMID 2242058
- [Background] Altman R, Alarcon G, Appelrouth D, Bloch D, Borenstein D, Brandt K, Brown C, Cooke TD, Daniel W, Feldman D, et al. The American College of Rheumatology criteria for the classification and reporting of osteoarthritis of the hip. Arthritis Rheum. 1991 May;34(5):505-14. doi: 10.1002/art.1780340502. PMID 2025304
- [Background] Al-Zahrani KS, Bakheit AM. A study of the gait characteristics of patients with chronic osteoarthritis of the knee. Disabil Rehabil. 2002 Mar 20;24(5):275-80. doi: 10.1080/09638280110087098. PMID 12004973
- [Background] Amin S, Baker K, Niu J, Clancy M, Goggins J, Guermazi A, Grigoryan M, Hunter DJ, Felson DT. Quadriceps strength and the risk of cartilage loss and symptom progression in knee osteoarthritis. Arthritis Rheum. 2009 Jan;60(1):189-98. doi: 10.1002/art.24182. PMID 19116936
- [Background] Arden N, Nevitt MC. Osteoarthritis: epidemiology. Best Pract Res Clin Rheumatol. 2006 Feb;20(1):3-25. doi: 10.1016/j.berh.2005.09.007. PMID 16483904
- [Background] Bellamy N, Buchanan WW, Goldsmith CH, Campbell J, Stitt LW. Validation study of WOMAC: a health status instrument for measuring clinically important patient relevant outcomes to antirheumatic drug therapy in patients with osteoarthritis of the hip or knee. J Rheumatol. 1988 Dec;15(12):1833-40. PMID 3068365
- [Background] Bennell KL, Hunt MA, Wrigley TV, Hunter DJ, McManus FJ, Hodges PW, Li L, Hinman RS. Hip strengthening reduces symptoms but not knee load in people with medial knee osteoarthritis and varus malalignment: a randomised controlled trial. Osteoarthritis Cartilage. 2010 May;18(5):621-8. doi: 10.1016/j.joca.2010.01.010. Epub 2010 Feb 6. PMID 20175973
- [Background] Boling MC, Bolgla LA, Mattacola CG, Uhl TL, Hosey RG. Outcomes of a weight-bearing rehabilitation program for patients diagnosed with patellofemoral pain syndrome. Arch Phys Med Rehabil. 2006 Nov;87(11):1428-35. doi: 10.1016/j.apmr.2006.07.264. PMID 17084115
- [Background] Cools AM, Vanderstukken F, Vereecken F, Duprez M, Heyman K, Goethals N, Johansson F. Eccentric and isometric shoulder rotator cuff strength testing using a hand-held dynamometer: reference values for overhead athletes. Knee Surg Sports Traumatol Arthrosc. 2016 Dec;24(12):3838-3847. doi: 10.1007/s00167-015-3755-9. Epub 2015 Aug 21. PMID 26294055
- [Background] Costa RA, Oliveira LM, Watanabe SH, Jones A, Natour J. Isokinetic assessment of the hip muscles in patients with osteoarthritis of the knee. Clinics (Sao Paulo). 2010;65(12):1253-9. doi: 10.1590/s1807-59322010001200006. PMID 21340212
- [Background] Culvenor AG, Wirth W, Roth M, Hunter DJ, Eckstein F. Predictive Capacity of Thigh Muscle Strength in Symptomatic and/or Radiographic Knee Osteoarthritis Progression: Data from the Foundation for the National Institutes of Health Osteoarthritis Biomarkers Consortium. Am J Phys Med Rehabil. 2016 Dec;95(12):931-938. doi: 10.1097/PHM.0000000000000534. PMID 27175558
- [Background] Eckstein F, Wirth W, Nevitt MC. Recent advances in osteoarthritis imaging--the osteoarthritis initiative. Nat Rev Rheumatol. 2012 Oct;8(10):622-30. doi: 10.1038/nrrheum.2012.113. Epub 2012 Jul 10. PMID 22782003
- [Background] Eckstein F, Hitzl W, Duryea J, Kent Kwoh C, Wirth W; OAI investigators. Baseline and longitudinal change in isometric muscle strength prior to radiographic progression in osteoarthritic and pre-osteoarthritic knees--data from the Osteoarthritis Initiative. Osteoarthritis Cartilage. 2013 May;21(5):682-90. doi: 10.1016/j.joca.2013.02.658. Epub 2013 Mar 6. PMID 23473978
- [Background] Farr JN, Going SB, Lohman TG, Rankin L, Kasle S, Cornett M, Cussler E. Physical activity levels in patients with early knee osteoarthritis measured by accelerometry. Arthritis Rheum. 2008 Sep 15;59(9):1229-36. doi: 10.1002/art.24007. PMID 18759320
- [Background] Ferber R, Bolgla L, Earl-Boehm JE, Emery C, Hamstra-Wright K. Strengthening of the hip and core versus knee muscles for the treatment of patellofemoral pain: a multicenter randomized controlled trial. J Athl Train. 2015 Apr;50(4):366-77. doi: 10.4085/1062-6050-49.3.70. Epub 2014 Nov 3. PMID 25365133
- [Background] Fukuda TY, Rossetto FM, Magalhaes E, Bryk FF, Lucareli PR, de Almeida Aparecida Carvalho N. Short-term effects of hip abductors and lateral rotators strengthening in females with patellofemoral pain syndrome: a randomized controlled clinical trial. J Orthop Sports Phys Ther. 2010 Nov;40(11):736-42. doi: 10.2519/jospt.2010.3246. PMID 21041965
- [Background] Fukuda TY, Melo WP, Zaffalon BM, Rossetto FM, Magalhaes E, Bryk FF, Martin RL. Hip posterolateral musculature strengthening in sedentary women with patellofemoral pain syndrome: a randomized controlled clinical trial with 1-year follow-up. J Orthop Sports Phys Ther. 2012 Oct;42(10):823-30. doi: 10.2519/jospt.2012.4184. Epub 2012 Aug 2. PMID 22951491
- [Background] Glass NA, Torner JC, Frey Law LA, Wang K, Yang T, Nevitt MC, Felson DT, Lewis CE, Segal NA. The relationship between quadriceps muscle weakness and worsening of knee pain in the MOST cohort: a 5-year longitudinal study. Osteoarthritis Cartilage. 2013 Sep;21(9):1154-9. doi: 10.1016/j.joca.2013.05.016. PMID 23973125
- [Background] Hinman RS, Hunt MA, Creaby MW, Wrigley TV, McManus FJ, Bennell KL. Hip muscle weakness in individuals with medial knee osteoarthritis. Arthritis Care Res (Hoboken). 2010 Aug;62(8):1190-3. doi: 10.1002/acr.20199. PMID 20704005
- [Background] Hott A, Liavaag S, Juel NG, Brox JI. Study protocol: a randomised controlled trial comparing the long term effects of isolated hip strengthening, quadriceps-based training and free physical activity for patellofemoral pain syndrome (anterior knee pain). BMC Musculoskelet Disord. 2015 Feb 25;16:40. doi: 10.1186/s12891-015-0493-6. PMID 25879452
- [Background] Hu B, Skou ST, Wise BL, Williams GN, Nevitt MC, Segal NA. Lower Quadriceps Rate of Force Development Is Associated With Worsening Physical Function in Adults With or at Risk for Knee Osteoarthritis: 36-Month Follow-Up Data From the Osteoarthritis Initiative. Arch Phys Med Rehabil. 2018 Jul;99(7):1352-1359. doi: 10.1016/j.apmr.2017.12.027. Epub 2018 Jan 31. PMID 29408538
- [Background] Hurd WJ, Morrey BF, Kaufman KR. The effects of anthropometric scaling parameters on normalized muscle strength in uninjured baseball pitchers. J Sport Rehabil. 2011 Aug;20(3):311-20. doi: 10.1123/jsr.20.3.311. PMID 21828383
- [Background] Ismail MM, Gamaleldein MH, Hassa KA. Closed kinetic chain exercises with or without additional hip strengthening exercises in management of patellofemoral pain syndrome: a randomized controlled trial. Eur J Phys Rehabil Med. 2013 Oct;49(5):687-98. Epub 2013 Jul 2. PMID 23820880
- [Background] KELLGREN JH, LAWRENCE JS. Radiological assessment of osteo-arthrosis. Ann Rheum Dis. 1957 Dec;16(4):494-502. doi: 10.1136/ard.16.4.494. No abstract available. PMID 13498604
- [Background] Kemnitz J, Wirth W, Eckstein F, Ruhdorfer A, Culvenor AG. Longitudinal change in thigh muscle strength prior to and concurrent with symptomatic and radiographic knee osteoarthritis progression: data from the Osteoarthritis Initiative. Osteoarthritis Cartilage. 2017 Oct;25(10):1633-1640. doi: 10.1016/j.joca.2017.07.003. Epub 2017 Jul 8. PMID 28698106
- [Background] Khayambashi K, Mohammadkhani Z, Ghaznavi K, Lyle MA, Powers CM. The effects of isolated hip abductor and external rotator muscle strengthening on pain, health status, and hip strength in females with patellofemoral pain: a randomized controlled trial. J Orthop Sports Phys Ther. 2012 Jan;42(1):22-9. doi: 10.2519/jospt.2012.3704. Epub 2011 Oct 25. PMID 22027216
- [Background] Liao CD, Huang YC, Lin LF, Huang SW, Liou TH. Body mass index and functional mobility outcome following early rehabilitation after a total knee replacement: a retrospective study in Taiwan. Arthritis Care Res (Hoboken). 2015 May;67(6):799-808. doi: 10.1002/acr.22474. PMID 25201765
- [Background] Martin HJ, Yule V, Syddall HE, Dennison EM, Cooper C, Aihie Sayer A. Is hand-held dynamometry useful for the measurement of quadriceps strength in older people? A comparison with the gold standard Bodex dynamometry. Gerontology. 2006;52(3):154-9. doi: 10.1159/000091824. PMID 16645295
- [Background] McNair PJ, Colvin M, Reid D. Predicting maximal strength of quadriceps from submaximal performance in individuals with knee joint osteoarthritis. Arthritis Care Res (Hoboken). 2011 Feb;63(2):216-22. doi: 10.1002/acr.20368. PMID 20890972
- [Background] Messier SP, Mihalko SL, Beavers DP, Nicklas BJ, DeVita P, Carr JJ, Hunter DJ, Williamson JD, Bennell KL, Guermazi A, Lyles M, Loeser RF. Strength Training for Arthritis Trial (START): design and rationale. BMC Musculoskelet Disord. 2013 Jul 15;14:208. doi: 10.1186/1471-2474-14-208. PMID 23855596
- [Background] Palmer K, Hebron C, Williams JM. A randomised trial into the effect of an isolated hip abductor strengthening programme and a functional motor control programme on knee kinematics and hip muscle strength. BMC Musculoskelet Disord. 2015 May 3;16:105. doi: 10.1186/s12891-015-0563-9. PMID 25935843
- [Background] Rikli RE, Jones CJ. Development and validation of criterion-referenced clinically relevant fitness standards for maintaining physical independence in later years. Gerontologist. 2013 Apr;53(2):255-67. doi: 10.1093/geront/gns071. Epub 2012 May 20. PMID 22613940
- [Background] Ringdahl E, Pandit S. Treatment of knee osteoarthritis. Am Fam Physician. 2011 Jun 1;83(11):1287-92. PMID 21661710
- [Background] Ruhdorfer A, Dannhauer T, Wirth W, Hitzl W, Kwoh CK, Guermazi A, Hunter DJ, Benichou O, Eckstein F; Osteoarthritis Initiative Investigators. Thigh muscle cross-sectional areas and strength in advanced versus early painful osteoarthritis: an exploratory between-knee, within-person comparison in osteoarthritis initiative participants. Arthritis Care Res (Hoboken). 2013 Jul;65(7):1034-42. doi: 10.1002/acr.21965. PMID 23401316
- [Background] Ruhdorfer A, Wirth W, Hitzl W, Nevitt M, Eckstein F; Osteoarthritis Initiative Investigators. Association of thigh muscle strength with knee symptoms and radiographic disease stage of osteoarthritis: data from the Osteoarthritis Initiative. Arthritis Care Res (Hoboken). 2014 Sep;66(9):1344-53. doi: 10.1002/acr.22317. PMID 24578353
- [Background] Ruhdorfer A, Wirth W, Eckstein F. Longitudinal Change in Thigh Muscle Strength Prior to and Concurrent With Minimum Clinically Important Worsening or Improvement in Knee Function: Data From the Osteoarthritis Initiative. Arthritis Rheumatol. 2016 Apr;68(4):826-36. doi: 10.1002/art.39484. PMID 26556499
- [Background] Schache MB, McClelland JA, Webster KE. Does the addition of hip strengthening exercises improve outcomes following total knee arthroplasty? A study protocol for a randomized trial. BMC Musculoskelet Disord. 2016 Jun 13;17:259. doi: 10.1186/s12891-016-1104-x. PMID 27295978
- [Background] Segal NA, Glass NA, Torner J, Yang M, Felson DT, Sharma L, Nevitt M, Lewis CE. Quadriceps weakness predicts risk for knee joint space narrowing in women in the MOST cohort. Osteoarthritis Cartilage. 2010 Jun;18(6):769-75. doi: 10.1016/j.joca.2010.02.002. Epub 2010 Feb 11. PMID 20188686
- [Background] Segal NA, Findlay C, Wang K, Torner JC, Nevitt MC. The longitudinal relationship between thigh muscle mass and the development of knee osteoarthritis. Osteoarthritis Cartilage. 2012 Dec;20(12):1534-40. doi: 10.1016/j.joca.2012.08.019. Epub 2012 Sep 3. PMID 22954456
- [Background] Sharma L, Dunlop DD, Cahue S, Song J, Hayes KW. Quadriceps strength and osteoarthritis progression in malaligned and lax knees. Ann Intern Med. 2003 Apr 15;138(8):613-9. doi: 10.7326/0003-4819-138-8-200304150-00006. PMID 12693882
- [Background] Skou ST, Simonsen O, Rasmussen S. Examination of muscle strength and pressure pain thresholds in knee osteoarthritis: test-retest reliability and agreement. J Geriatr Phys Ther. 2015 Jul-Sep;38(3):141-7. doi: 10.1519/JPT.0000000000000028. PMID 25594517
- [Background] Sled EA, Khoja L, Deluzio KJ, Olney SJ, Culham EG. Effect of a home program of hip abductor exercises on knee joint loading, strength, function, and pain in people with knee osteoarthritis: a clinical trial. Phys Ther. 2010 Jun;90(6):895-904. doi: 10.2522/ptj.20090294. Epub 2010 Apr 8. PMID 20378679
- [Background] Xie Y, Zhang C, Jiang W, Huang J, Xu L, Pang G, Tang H, Chen R, Yu J, Guo S, Xu F, Wang J. Quadriceps combined with hip abductor strengthening versus quadriceps strengthening in treating knee osteoarthritis: a study protocol for a randomized controlled trial. BMC Musculoskelet Disord. 2018 May 15;19(1):147. doi: 10.1186/s12891-018-2041-7. PMID 29764409
- [Background] Zeni JA Jr, Axe MJ, Snyder-Mackler L. Clinical predictors of elective total joint replacement in persons with end-stage knee osteoarthritis. BMC Musculoskelet Disord. 2010 May 6;11:86. doi: 10.1186/1471-2474-11-86. PMID 20459622